CLINICAL TRIAL: NCT05990569
Title: A Randomized Comparative Study of Pudendal Nerve Block With Bupivacaine Alone and Bupivacaine With Methylene Blue for Postoperative Analgesia in Perianal Surgery
Brief Title: Pudendal Nerve Block With Bupivacaine Alone and Bupivacaine With Methylene Blue for Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Saurav Raj Khatiwada, Resident Doctor, Nepal Mediciti Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRC-RP-2079/80-04
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Hemorrhoids; Anal Fissure and Fistula; Perianal Abscess; Perianal Fistula; Pilonidal Sinus; Perianal Skin Tags
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano; Fistula; Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Bupivacaine
  Interventions: Other: Ultrasound guided Pudendal nerve block
- Arm B (Experimental): Bupivacaine with methylene blue
  Interventions: Other: Ultrasound guided Pudendal nerve block

INTERVENTIONS:
Other: Ultrasound guided Pudendal nerve block — Ultrasound guided bilateral pudendal nerve block

SUMMARY:
Study Description:

The goal of this clinical trial is to compare the duration of postoperative pain relief achieved with two different approaches to pudendal nerve block in patients undergoing elective perianal surgery. The main question this study aims to answer is whether adding Methylene Blue to Bupivacaine pudendal nerve block can prolong postoperative analgesia compared to using Bupivacaine alone.

Participants in this study will be individuals with ASA I and II physical status undergoing elective perianal surgery under spinal anesthesia. They will be randomly assigned to one of two groups:

1. Group A (Case Group): Participants will receive a pudendal nerve block with Bupivacaine combined with Methylene Blue.
2. Group B (Control Group): Participants will receive a pudendal nerve block with Bupivacaine alone.

The pudendal nerve block will be performed using ultrasound guidance at the level of the ischial spine. The needle tip will be positioned between the Sacro tuberous and sacrospinous ligaments to inject the local anesthetic or the local anesthetic combined with Methylene Blue.

Throughout the study, the researchers will monitor the time to the first rescue analgesic, assess pain levels using the Numeric Rating Scale at various time intervals (2, 6, 24, 48 hours, and 7 days), and observe for any side effects or complications related to the intervention.

Participants will be closely observed after surgery to assess their pain levels and analgesic requirements. The researchers will also evaluate patient satisfaction using the Likert scale.

By comparing the outcomes between the two groups, the study aims to determine if the addition of Methylene Blue to Bupivacaine pudendal nerve block provides superior postoperative analgesia in perianal surgery patients. This information will contribute to the understanding of effective pain management strategies for individuals undergoing perianal surgical procedures and potentially reduce the need for opioids and improve patient outcomes.

DETAILED DESCRIPTION:
Study Description:

The aim of this randomized comparative study is to investigate the effectiveness of two different approaches to postoperative analgesia in patients undergoing perianal surgery. The study will compare the use of Bupivacaine alone with Bupivacaine combined with Methylene Blue in a pudendal nerve block.

Perianal surgical procedures, such as abscess drainage, fistulectomy, and hemorrhoidectomy, can cause significant postoperative pain. The goal of this study is to find a more effective and prolonged method of pain relief to improve patient comfort and reduce the need for opioids.

Participants in this study will be individuals scheduled for elective perianal surgery and classified as ASA I and II. They will be randomly assigned to one of two groups:

1. Group A: Participants will receive a pudendal nerve block with Bupivacaine and Methylene Blue.
2. Group B: Participants will receive a pudendal nerve block with Bupivacaine alone.

The pudendal nerve block will be performed under ultrasound guidance at the ischial spine level. The needle will be accurately placed between the Sacro tuberous and sacrospinous ligaments for precise injection of the local anesthetic or the local anesthetic combined with Methylene Blue.

Throughout the study, the researchers will closely monitor the participants to assess the time to the first rescue analgesic and pain levels using the Numeric Rating Scale at specific time intervals (2, 6, 24, 48 hours, and 7 days). Additionally, any side effects, allergies, itching, hematoma, infection, or complications like loss of anal sphincter function will be recorded.

Patient satisfaction will also be evaluated using the Likert scale to determine the perceived effectiveness of the different approaches to postoperative analgesia.

By comparing the outcomes between the two groups, this study aims to determine whether the addition of Methylene Blue to Bupivacaine in a pudendal nerve block can prolong postoperative analgesia in patients undergoing perianal surgery. The findings from this study may contribute valuable insights into improving pain management strategies and enhancing the overall recovery experience for patients undergoing perianal surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients of ASA I and II undergoing elective perianal surgery under spinal anesthesia

Exclusion Criteria:

1. Patient's refusal
2. Patient with a history of allergy to the local anesthetic or Methylene blue
3. Bleeding diathesis or coagulopathy
4. Extensive infection at the site of injection
5. Pregnancy and lactating mother
6. Spinal abnormality
7. Patients with neurological deficit

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Time to the first rescue analgesic administration (in minutes) in the two study groups | 48 hours
  We will compare the time at which patients in either group will demand rescue analgesic
Patient satisfaction assessed using the Likert scale after receiving Bupivacaine pudendal nerve block with or without Methylene Blue. | Seven days
  We will ask the patient to select one of the following satisfaction scores:
  Very satisfied Moderately satisfied Neither satisfied nor dissatisfied Moderately dissatisfied Very dissatisfied

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) score for pain intensity at different time intervals | Seven days
  Numeric Rating Scale (NRS) score for pain intensity will be measured at different time intervals (at 2, 6, 24, 48 hours, and 7 days) after surgery in both study groups.
Complications | seven days
  Incidence of complications related to the pudendal nerve block procedure, such as hematoma, infection, and allergic reactions will be captured when it is detected or at the end of seventh postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Pragati Koirala, MD, Principal Investigator — Nepal Mediciti
Locations (1):
- Nepal Mediciti Hospital, Lalitpur, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imbelloni LE, Vieira EM, Gouveia MA, Netinho JG, Spirandelli LD, Cordeiro JA. Pudendal block with bupivacaine for postoperative pain relief. Dis Colon Rectum. 2007 Oct;50(10):1656-61. doi: 10.1007/s10350-007-0216-7. PMID 17701375
- [Background] Sim HL, Tan KY. Randomized single-blind clinical trial of intradermal methylene blue on pain reduction after open diathermy haemorrhoidectomy. Colorectal Dis. 2014 Aug;16(8):O283-7. doi: 10.1111/codi.12587. PMID 24506265
- [Background] Naja Z, Ziade MF, Lonnqvist PA. Nerve stimulator guided pudendal nerve block decreases posthemorrhoidectomy pain. Can J Anaesth. 2005 Jan;52(1):62-8. doi: 10.1007/BF03018582. PMID 15625258
- [Background] Kunitake H, Poylin V. Complications Following Anorectal Surgery. Clin Colon Rectal Surg. 2016 Mar;29(1):14-21. doi: 10.1055/s-0035-1568145. PMID 26929747
- [Background] Ceulemans A, De Looze D, Van de Putte D, Stiers E, Coppens M. High post-operative pain scores despite multimodal analgesia in ambulatory anorectal surgery: a prospective cohort study. Acta Chir Belg. 2019 Aug;119(4):224-230. doi: 10.1080/00015458.2018.1500802. Epub 2018 Sep 7. PMID 30189793
- [Background] Garimella V, Cellini C. Postoperative pain control. Clin Colon Rectal Surg. 2013 Sep;26(3):191-6. doi: 10.1055/s-0033-1351138. PMID 24436674
- [Background] Abdi S, Shenouda P, Patel N, Saini B, Bharat Y, Calvillo O. A novel technique for pudendal nerve block. Pain Physician. 2004 Jul;7(3):319-22. PMID 16858468
- [Background] Ginimuge PR, Jyothi SD. Methylene blue: revisited. J Anaesthesiol Clin Pharmacol. 2010 Oct;26(4):517-20. No abstract available. PMID 21547182
- [Background] Lee SW, Han HC. Methylene Blue Application to Lessen Pain: Its Analgesic Effect and Mechanism. Front Neurosci. 2021 May 17;15:663650. doi: 10.3389/fnins.2021.663650. eCollection 2021. PMID 34079436
- [Background] Steen CJ, Lam D, Chandra R, Chua JYJ, An V, Keck JO. Pudendal Nerve Block for Posthemorrhoidectomy Pain: A Prospective, Single-Blinded Randomized Control Trial. Dis Colon Rectum. 2022 Apr 1;65(4):546-551. doi: 10.1097/DCR.0000000000002293. PMID 34759239